CLINICAL TRIAL: NCT02701894
Title: The Effect of Alpha-Linolenic Acid on Glycemic Control in Participants With Type 2 Diabetes
Brief Title: ALA on Glycemic Control in T2DM Participants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Vladimir Vuksan, Research Scientist & Professor, Unity Health Toronto
Other Study IDs: ALA and GC in T2D
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alpha-Linolenic Acid

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Alpha-Linolenic Acid — Meta-Analysis of Randomized Controlled Trials
  Other Names: ALA

SUMMARY:
With the emerging worldwide epidemic of type 2 diabetes, dietary recommendations to improve diabetes management have been emphasized in the scientific community. Particular attention has been drawn to various benefits of replacing saturated fatty acids with unsaturated fatty acids. Alpha-linolenic acid, the only omega-3 fatty acid that is from plant sources, has been suggested by animal and cell studies to play a beneficial role in regulating blood glucose levels. However, human studies have been more inconsistent with their findings. The focus of this project is to investigate the evidence in the context of ALA and blood glucose parameters in participants with type 2 diabetes by conducting a systematic review and meta-analysis of randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Controlled, randomized, clinical trials
* Trials greater than one month
* Focusing on ALA and T2DM participants
* Viable endpoint data

Exclusion Criteria:

* Non-human studies
* Non-random treatment allocation
* Less than 1 month
* Lack of suitable control
* Lack of endpoint data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 2 diabetes mellitus.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 1 month

SECONDARY OUTCOMES:
Fructosamine | 1 month
Fasting Blood Glucose | 1 month
Fasting Blood Insulin | 1 month
Glycated Albumin | 1 month
HOMA- IR | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto